CLINICAL TRIAL: NCT04596553
Title: The Effects of Essential and Non-Essential Amino Acids on Post-Exercise Muscle Collagen Synthesis in Young Men: a Randomized Controlled Trial
Brief Title: Effects of Essential and Non-Essential Amino Acids on Post-Exercise Muscle Collagen Synthesis in Young Men
Acronym: PECS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Cameron Mitchell, Assistant Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: H20-00943
Record Dates: First submitted 2020-09-28; First posted 2020-10-22 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Skeletal Muscle; Extracellular Matrix; Amino Acids Metabolism; Exercise; Dietary Supplements
Keywords: Muscle Collagen Turnover; Myofibrillar Protein Synthesis; Extracellular Matrix; Anabolism Signaling; Resistance Exercise; Skeletal Muscle; Bone Turnover
MeSH Terms: conditions — Motor Activity | interventions — Amino Acids, Essential

STUDY DESIGN:
Intervention Model Description: - Double-blinded, randomized controlled, parallel design study, with 3 treatment groups (placebo, collagen peptide, and essential amino acid)
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Essential Amino Acid (Active Comparator): Participants will consume 1 dose of: 15 g crystalline essential amino acid supplement (Pure Encapsulation Essential Aminos 180) + 80 ml (48 mg) Vitamin C (Ribena Blackcurrant) + 250 ml water
  Interventions: Dietary Supplement: Essential Amino Acid
- Collagen Peptide (Active Comparator): Participants will consume 1 dose of: 15g collagen peptide (Gelita TENDOFORTE) + 80 ml (48 mg) Vitamin C (Ribena Blackcurrant) + 250 ml water
  Interventions: Dietary Supplement: Collagen Peptide
- Maltodextrin Placebo (Placebo Comparator): Participants will consume 1 dose of:15 g maltodextrin (Canadian Protein Maltodextrin) + 80 ml (48 mg) Vitamin C (Ribena Blackcurrant) + 250 ml water
  Interventions: Dietary Supplement: Maltodextrin Placebo

INTERVENTIONS:
Dietary Supplement: Essential Amino Acid — Immediately following the exercise intervention participants will consume their assigned essential amino acid supplement
  Arms: Essential Amino Acid
Dietary Supplement: Collagen Peptide — Immediately following the exercise intervention participants will consume their assigned collagen peptide supplement
  Arms: Collagen Peptide
Dietary Supplement: Maltodextrin Placebo — Immediately following the exercise intervention participants will consume their assigned maltodextrin supplement
  Arms: Maltodextrin Placebo

SUMMARY:
The purpose of this study is to assess which amino acids are affecting acute muscle collagen synthesis in response to supplementation and exercise.

DETAILED DESCRIPTION:
This is a double-blinded, randomized controlled, parallel design study, with 3 treatment groups (placebo, collagen peptide, and essential amino acid). The study will involve 3 visits: a baseline testing/familiarization session, and 2 exercise trials which will include muscle biopsies, blood draws, and the infusion of a tracer isotope in order to measure muscle protein synthesis.

ELIGIBILITY:
Inclusion Criteria:

* Can fluently read and write in English
* Male
* 18 - 35 years

Exclusion Criteria:

* Diabetes, cardiovascular disease, or current pharmaceutical therapy
* Medical conditions impacting ability to undertake strenuous physical activity
* Lower body resistance training in the previous 6 months
* BMI > 30
* Currently smoking with cigarettes
* Allergy to any study supplements
* Currently taking any protein, amino acid, or collagen supplement
* Participate in greater than 2 hours of weekly vigorous exercise

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2021-01-25 (Actual); Primary Completion 2022-02-13 (Actual); Study Completion 2022-02-13 (Actual)

PRIMARY OUTCOMES:
Fractional synthetic rate (change over time) of Myofibrillar Protein Synthesis | 0 - 4 hours post-exercise
  Fraction of the myofibrillar enriched protein from muscle biopsy per unit time.
Fractional synthetic rate (change over time) of Myofibrillar Protein Synthesis | 0 - 2 hours post-exercise
  Fraction of the myofibrillar enriched protein from muscle biopsy per unit time.
Fractional synthetic rate (change over time) of Myofibrillar Protein Synthesis | 2 - 4 hours post-exercise
  Fraction of the myofibrillar enriched protein from muscle biopsy per unit time.
Fractional synthetic rate (change over time) Muscle Collagen Synthesis | 0 - 4 hours post-exercise
  Fraction of the intramuscular collagen enriched protein from muscle biopsy per unit time.
Fractional synthetic rate (change over time) Muscle Collagen Synthesis | 0 - 2 hours post-exercise
  Fraction of the intramuscular collagen enriched protein from muscle biopsy per unit time.
Fractional synthetic rate (change over time) Muscle Collagen Synthesis | 2 - 4 hours post-exercise
  Fraction of the intramuscular collagen enriched protein from muscle biopsy per unit time.
Pro-Collagen Type I N-Propeptide (PINP) | 1 hour prior to exercise
  Osteoblastic marker of bone collagen synthesis
Pro-Collagen Type I N-Propeptide (PINP) | 4 hours post exercise
  Osteoblastic marker of bone collagen synthesis

SECONDARY OUTCOMES:
Plasma Amino Acids Response to Supplementation | 0 - 4 hours post-exercise
  Amino acid plasma concentrations
Muscle mechanistic target of rapamycin Pathway Activation | 0 - 4 hours post-exercise
  Measuring the fold change in enzymes associated with the anabolic signalling of the mTOR pathway (e.g. phosphoinositide 3-kinases (PI3k), protein kinase B (Akt))
PCR Gene Expression of Muscle Collagen Genes (Types I, III, IV) | 0 - 4 hours post-exercise
  Measuring the fold change when the collagen genes of interest become detectable in the PCR analysis
Pro-Collagen Type III N-Propeptide (PIIINP) | 1 hour prior to exercise
  Marker of collagen synthesis
Pro-Collagen Type III N-Propeptide (PIIINP) | 4 hours post exercise
  Marker of collagen synthesis

CONTACTS AND LOCATIONS:
Overall Officials: Cameron Mitchell, PhD, Principal Investigator — University of British Columbia
Locations (1):
- Chan Gunn Pavilion, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shaw G, Lee-Barthel A, Ross ML, Wang B, Baar K. Vitamin C-enriched gelatin supplementation before intermittent activity augments collagen synthesis. Am J Clin Nutr. 2017 Jan;105(1):136-143. doi: 10.3945/ajcn.116.138594. Epub 2016 Nov 16. PMID 27852613
- [Background] Holm L, Rahbek SK, Farup J, Vendelbo MH, Vissing K. Contraction mode and whey protein intake affect the synthesis rate of intramuscular connective tissue. Muscle Nerve. 2017 Jan;55(1):128-130. doi: 10.1002/mus.25398. Epub 2016 Sep 26. PMID 27603578
- [Background] Frontera WR, Ochala J. Skeletal muscle: a brief review of structure and function. Calcif Tissue Int. 2015 Mar;96(3):183-95. doi: 10.1007/s00223-014-9915-y. Epub 2014 Oct 8. PMID 25294644
- [Background] Egerman MA, Glass DJ. Signaling pathways controlling skeletal muscle mass. Crit Rev Biochem Mol Biol. 2014 Jan-Feb;49(1):59-68. doi: 10.3109/10409238.2013.857291. Epub 2013 Nov 18. PMID 24237131
- [Background] Holm L, van Hall G, Rose AJ, Miller BF, Doessing S, Richter EA, Kjaer M. Contraction intensity and feeding affect collagen and myofibrillar protein synthesis rates differently in human skeletal muscle. Am J Physiol Endocrinol Metab. 2010 Feb;298(2):E257-69. doi: 10.1152/ajpendo.00609.2009. Epub 2009 Nov 10. PMID 19903866
- [Background] Alcock RD, Shaw GC, Tee N, Burke LM. Plasma Amino Acid Concentrations After the Ingestion of Dairy and Collagen Proteins, in Healthy Active Males. Front Nutr. 2019 Oct 15;6:163. doi: 10.3389/fnut.2019.00163. eCollection 2019. PMID 31681789
- [Background] Miller BF, Olesen JL, Hansen M, Dossing S, Crameri RM, Welling RJ, Langberg H, Flyvbjerg A, Kjaer M, Babraj JA, Smith K, Rennie MJ. Coordinated collagen and muscle protein synthesis in human patella tendon and quadriceps muscle after exercise. J Physiol. 2005 Sep 15;567(Pt 3):1021-33. doi: 10.1113/jphysiol.2005.093690. Epub 2005 Jul 7. PMID 16002437